CLINICAL TRIAL: NCT00746070
Title: Postoperative Cardiovascular Index Change of Primary Aldosteronism
Acronym: TAIPAI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: VinCent Wu, Nation Taiwan University Hospital
Other Study IDs: 200611031R
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-04

CONDITIONS: Aldosteronism
Keywords: cardiovascular disease, endothelium function, aldosterone
MeSH Terms: conditions — Hyperaldosteronism; Cardiovascular Diseases | interventions — Spironolactone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A, primary aldosteronism: patients approved to be aldosteronism
  Interventions: Other: with the clinical treatment ( ex adrenalectomy or spironolactone
- B, essential hypertension: patients approved to be essential hypertension

INTERVENTIONS:
Other: with the clinical treatment ( ex adrenalectomy or spironolactone — with the clinical observational study
  Groups: A, primary aldosteronism

SUMMARY:
Primary aldosteronism (PA), characterized by an inappropriate production of aldosterone, is far more common than is usually perceived. The overall prevalence of PA is 11.2% of the newly diagnosed hypertensive patients and 4.8% was curable aldosterone producing adenoma (APA), and adrenalectomy is considered the treatment of choice for APA. The potential curability and prevention of excess cardiovascular damage and events also underscores the need to develop accurate strategies for the timely diagnosis of APA.This study aimed to determine the effects of endothelium function change ( PWV, progenitor cell,..) before and post-adrenalectomy or taking spironolactone in patients with aldosteronism. Autonomous elevated aldosterone will increase the glomerular filtration rate and renal damage in patients with primary aldosteronism (PA). But clinical evidence of the role of endothelium function on post-adrenalectomy or taking spirolactone is still limited.

DETAILED DESCRIPTION:
Aldosterone has rapid nongenomic effects in the human vasculature. Aldosterone has been claimed to lead to endothelial dysfunction, a condition related to development of cardiovascular disorders and to poor prognosis. However, studies of aldosterone effects on endothelial function led to discrepant findings, which may be related, at least in part, to inhomogeneity of the populations studied. Thus, studies in healthy subjects showed no detrimental effects of aldosterone on endothelial function and no positive effect of aldosterone inhibition, whereas populations with established cardiovascular diseases showed negative effects of aldosterone and positive effects of spironolactone therapy. Still, other factors may be of importance as effects of aldosterone on endothelial function are not homogenous even in a healthy population. Dosages of aldosterone, concomitant drug use, as well as the vascular bed investigated may influence the effects observed.

Furthermore, little is known about chronic endothelial effects of aldosterone that could indicate a primary and direct role of aldosterone in development of cardiovascular diseases. In patients with hyperaldosteronism diminished flow-mediated dilation was found, indicating impaired endothelial function compared with hypertensive patients without elevated aldosterone. However, it is not known whether these results represent endothelial dysfunction as the result of a direct aldosterone effect on the vasculature or a secondary effect attributable to more substantial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* aldosteronism with hyperaldosterone
* older than 18 year of age
* completed the informed consent

Exclusion Criteria:

* pregnancy
* bed-ridden
* could not do MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: aldosteronism Patients enrolled from initial screening test and recorded in the Taiwan Primary Aldosteornism Investigation (TAIPAI) database. The database was constructed for quality assurance since 2003 in one medical center (National Taiwan University Hospital, Taipei, Taiwan) and its three branch hospitals in different cities (National Taiwan University Hospital Yun-Lin branch, Yun-Lin, southern Taiwan; Far-Eastern Memorial Hospital, Taipei; Tao-Yuan General Hospital, Tao-Yuan, middle Taiwan). All patients with intention to confirm and requiring suppression test or adrenal venous sampling were recruited and data were prospectively collected.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Change of fibrosis and endothelium parameter | post operation or taking spirolactone 4m, 12m

SECONDARY OUTCOMES:
Cardiovascular events | post operation or taking spirolactone for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Hun Lin, MD, Study Chair — NTUH

REFERENCES:
- [Background] Wu VC, Chueh SC, Chang HW, Lin WC, Liu KL, Li HY, Lin YH, Wu KD, Hsieh BS. Bilateral aldosterone-producing adenomas: differentiation from bilateral adrenal hyperplasia. QJM. 2008 Jan;101(1):13-22. doi: 10.1093/qjmed/hcm101. PMID 18203722
- [Background] Chang HW, Wu VC, Huang CY, Huang HY, Chen YM, Chu TS, Wu KD, Hsieh BS. D4 dopamine receptor enhances angiotensin II-stimulated aldosterone secretion through PKC-epsilon and calcium signaling. Am J Physiol Endocrinol Metab. 2008 Mar;294(3):E622-9. doi: 10.1152/ajpendo.00657.2007. Epub 2008 Jan 2. PMID 18171914
- [Background] Chang HW, Chu TS, Huang HY, Chueh SC, Wu VC, Chen YM, Hsieh BS, Wu KD. Down-regulation of D2 dopamine receptor and increased protein kinase Cmu phosphorylation in aldosterone-producing adenoma play roles in aldosterone overproduction. J Clin Endocrinol Metab. 2007 May;92(5):1863-70. doi: 10.1210/jc.2006-2338. Epub 2007 Feb 13. PMID 17299068
- [Derived] Wu CH, Yang YW, Hung SC, Tsai YC, Hu YH, Lin YH, Chu TS, Wu KD, Wu VC. Effect of Treatment on Body Fluid in Patients with Unilateral Aldosterone Producing Adenoma: Adrenalectomy versus Spironolactone. Sci Rep. 2015 Oct 19;5:15297. doi: 10.1038/srep15297. PMID 26477337